CLINICAL TRIAL: NCT02628184
Title: A Case Study of a Maternity Service Development Programme and Its Influence on Inter-agency Collaboration
Brief Title: A Case Study of a Maternity Service Development Programme
Status: Completed | Type: Observational
Sponsor: University of Southampton (Other)
Responsible Party: Sponsor
Other Study IDs: 13383; 170005 (Other: NHS)
Record Dates: First submitted 2015-07-14; First posted 2015-12-11 (Estimated); Last update posted 2021-06-16 (Actual); Status verified 2021-06

CONDITIONS: Collaboration

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Maternity Services Development Programme — The Maternity Services Development Programme was implemented to improve care for local families (service users) involved with maternity services. The aim was to improve care during the early stages of a family's development and to establish foundations for long-term well-being. One aspect of the programme worked to improve the delivery of care by facilitating collaboration and joint-planning between service providers. The programme uses local city Children's Centres to co-locate services (different agencies or professionals who are working within the same locality). The aim of co-location was to promote stronger collaboration between maternity services and other service provider agencies to develop stronger partnerships, and to help identify those who are (or who may become) vulnerable.
  Other Names: The Nurture Programme

SUMMARY:
BACKGROUND: In 2011 a Maternity Services Development Programme was implemented in a South of England city, to promote effective collaborative working between maternity services (midwives) and other service providers (health visitors, social workers, specialist services etc.) by co-locating services in local childrens centres. The progamme ultimately aimed to improve care for local service users (women and their families), especially those considered vulnerable. Implemented changes were based on evidence that suggests poor collaborative working contributes to poorer outcomes. RATIONALE: To explore the impact of the programme on local service providers, and by association service user care. AIM: To explore a localised Maternity Services Development Programme, identifying how inter- agency collaborative working occurs, and the service providers perceived benefits and challenges on collaboration, and by association service user care. METHODOLOGY: The proposed research uses a case study approach to collect and analyse predominantly qualitative data, and some quantitative data. Data will be collected using observation episodes (e.g. participant meetings) to observe collaboration, and interviews to explore these experiences. Additionally documents will be analysed to observe documented evidence of collaborative practice. Pre-existing statistical data will also be used to highlight changes in indicators of service user well being since the implementation of the Maternity Services Development Programme. PARTICIPANTS: A cross-section of service providers (no service users) working in or with maternity services from 4 of 9 city Children Centre's. FINDINGS: No current findings, data collection expected to start September 2015.

DETAILED DESCRIPTION:
In 2011 a Maternity Services Development Programme (MSDP) was implemented in one South of England city. The programme aimed to promote effective collaborative working between maternity services (midwives) and other service providers (health visitors, social workers, Children Centre staff, specialist and volunteer services) to improve outcomes for service users (women and families). The MSDP utilised local Children's Centres, which provide community focused family support, to co-locate maternity services and other service providers. The rationale to improve collaborative working is supported by evidence suggesting poor collaborative working contributes to poorer outcomes (Laming Report 2003; Marmot Review 2010). Therefore programmes such as the MSDP could potentially improve short and long-term outcomes for those accessing maternity services.

The proposed research uses a case study approach to collect and analyse predominantly qualitative data, and some quantitative data. This method will allow for analysis of the MSDP and understanding of its influence on maternity services and collaboration, and will aim to illuminate perceived strengths and challenges of the MSDP evident to services providers. Data will be collected using observation episodes (e.g. participant meetings) to observe collaboration, and interviews to explore experiences. Additionally documents will be analysed to observe documented evidence of collaborative practice. Pre-existing statistical data will also be used to highlight changes in indicators of service user well-being since the implementation of the MSDP.

The research will recruit a cross-section of service providers (no service users) that work in or with maternity services from four of the nine city Children Centres. Invitation letters will be circulated to potential participants through participating Children Centre management, where they will be invited to participate in the observation and interview data collection activities. They will then be able to select the extent of their participation.

ELIGIBILITY:
The inclusion criteria for this study is:

* Service providers working in, or from a local city Children's Centre (this may be in a practice base or working in the community);
* Service providers working in, or with maternity services;
* Service providers caring for families with women who are pregnant, or under the remit of maternity services (typically up to and including 6 weeks post-natally).

The exclusion criteria for this study is:

* Service providers caring for families with women no longer under the remit of maternity services (typically over 6 weeks post-natally).
* Service users (all women and families who use maternity services, inclusive of those considered vulnerable - this may be inclusive of some volunteer organisations who also provide services within children's centres).

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Service provider practitioners that have been influenced by the implementation of the Maternity Services Development Programme (including, Children Centre Staff and Practitioners (Centre Lead Practitioner/Manager, Family and Child practitioner and Frontline Receptionist), Midwives, Health Visitors, Social Workers and Additional Professional Practitioners (Nurture Practitioner, Parenting Practitioner and Early Years Teacher). Volunteer agencies have been excluded as many local groups are made up from community service users.
Sampling Method: Probability Sample
Enrollment: 19 (Actual)
Dates: Start 2016-01; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Perceived benefits or challenges of collaborative working | 2 Years

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Cluett, Study Director — University of Southampton; Jane March-McDonald, Study Director — University of Southampton
Locations (4):
- United Kingdom (4):
  - Buckland Children's Centre, Portsmouth, Hampshire
  - Mitlon Park Children's Centre, Portsmouth, Hampshire
  - Somerstown Children's Centre, Portsmouth, Hampshire
  - Paulsgrove Children's Centre, Portsmouth, Hampshire